CLINICAL TRIAL: NCT05252559
Title: Effect of Modified Ultrafiltration on Whole Blood Coagulation in Cardiac Surgery With Cardiopulmonary Bypass: Retrospective Analysis
Brief Title: Ultrafiltration on Coagulation Performance in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Tae-Yop Kim, MD PhD, Professor of Anesthesiology, Konkuk University Medical Center
Other Study IDs: 2019-05-008
Record Dates: First submitted 2022-01-25; First posted 2022-02-23 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Cardiac Valve Disease
Keywords: ultrafiltration; cardiac valve disease; viscoelastic test; cardiopulmonary bypass
MeSH Terms: conditions — Heart Valve Diseases | interventions — Ultrafiltration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: ultrafiltration — In cardiac surgery patients, ultrafiltration is usually applied to reduce free water and concentrate all blood components before weaning from cardiopulmonary bypass
Diagnostic Test: maximal clot firmness in EXTEM assay of ROTEM test — before and after applying ultrafiltration, arterial blood sample underwent EXTEM and FIBTEM assays of rotational thromboelastometry

SUMMARY:
In cardiac surgery patients with CPB-induced dilutional coagulopathy, ultrafiltration (UF) was applied to reduce free water and concentrate all blood components before the weaning from CPB. The impact of UF on the clot strength is determined by analyzing the changes of maximal clot formation in EXTEM assay (MCF-EXTEM) in the ROTEM test in patients who underwent elective cardiac valve surgery in KUMC.

DETAILED DESCRIPTION:
In cardiac surgery patients, ultrafiltration (UF) was applied to reduce free water and concentrate all blood components during cardiopulmonary bypass (CPB). Concentrating plasma substrate of UF would be beneficial in attenuating CPB-induced dilutional coagulopathy. This study was to investigate whether MUF affected viscoelastic profiles during CPB for cardiac surgery.

Patients who underwent elective cardiac surgery and MUF at the end of CPB during January 2019-December 2021 are recruited. Using the patients' electronic medical records, the values of maximum clot firmness of EXTEM assay (MCF-EXTEM) of rotational thromboelastometry (ROTEM) test before and after applying MUF are retrospectively analyzed.

As the primary measure, we determine the changes of MCF-EXTEM after applying MUF. With an assumption that MUF increased MCF-EXTEM, the receiver operating characteristic (ROC) analysis is applied to MCF-EXTEM change. The area under the ROC curve is determined and the cut-off value is estimated with specificity and sensitivity in Youden's J statistics. The change of MCF-EXTEM in patients who show MCF-EXTEM less than the cut-off value is analyzed. The changes of hematocrit (Hct) before and after applying MUF is also determined.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent cardiac surgery during Jan 2019-Dec 2021
* Patients underwent moderate hypothermic CPB
* Patients underwent ultrafiltration during CPB
* Patients underwent ROTEM tests (EXTEM assays and FIBTEM assay) before and after applying ultrafiltration

Exclusion Criteria:

* Patients underwent packed RBC transfusion > 3 units during CPB
* patients underwent ultrafiltration but the removed free water was < 250 ml
* Patients underwent deep hypothermia

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients underwent elective cardiac valve surgery with moderate hypothermic CPB and ultrafiltration
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
maximal clot firmness (MCF) of EXTEM assay | 30 minute after the completion of ultrafiltration
  change of MCF-EXTEM assay

SECONDARY OUTCOMES:
cut-off value of MCF-EXTEM to be improved by ultrafiltration | 30 minute after the completion of ultrafiltration
  To estimate the cut-off value of MCF-EXTEM which can be increased by applying ultrafiltration
maximal clot firmness (MCF) of EXTEM assay to be improved by ultrafiltration | 30 minute after the completion of ultrafiltration
  change of MCF-EXTEM by applying ultrafiltration in patients with reduced MCF-EXTEM before applying ultrafiltration (MCF-EXTEM < the estimated cut-off value)
maximal clot firmness (MCF) of EXTEM assay not to be improved by ultrafiltration | 30 minute after the completion of ultrafiltration
  change of MCF-EXTEM by applying ultrafiltration in patients with reduced MCF-EXTEM before applying ultrafiltration (MCF-EXTEM > the estimated cut-off value)

CONTACTS AND LOCATIONS:
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No